CLINICAL TRIAL: NCT06020729
Title: Effects of Occlusion Training on Speed and Physical Performance in Hockey Players
Brief Title: Effects of Occlusion Training on Hockey Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0403
Record Dates: First submitted 2023-04-18; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Sports Physical Therapy
Keywords: field hockey, muscle hypertrophy, occlusion training, power

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusion Training (Experimental)
  Interventions: Other: Occlusion Training
- General exercises without occlusion (Active Comparator)
  Interventions: Other: General Exercises without occlusion training

INTERVENTIONS:
Other: General Exercises without occlusion training — General Exercises as bench press, squats , maximum sprint, leg power without occlusion training
  Arms: General exercises without occlusion
Other: Occlusion Training — In experimental sessions players will perform with occlusion training which is blood flow resistance training, 4 times a week for 4 weeks with 5 sets of 5 repetitions and then assessed pre-training and post-training values with assessment tools bench press, leg squat, leg power, maximum sprint time.This training will also improve and increase muscular strength as well as speed and physical performance in players.
  Arms: Occlusion Training

SUMMARY:
Occlusion training is simply a way of restricting blood flow in the veins of a working muscle in hopes to kick-start some larger gains in muscle size and strength. Occlusion training performed during hockey training on speed and physical performance of hockey players. This training also known as blood flow restriction training, can be defined as the training of muscles while limiting blood flow to the muscles and typically done by performing high intensity, low weight, lifts while using some form of tourniquet or band to limit blood supply to limb being trained.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and total sample size of both groups will be 18 and calculated through non-probability sampling technique and the players will allocate into two groups, control group and experimental group, per group sample size is 9. Each will perform the session for occlusion training. Before and after training sessions players completed a series of test to assess their speed and physical performance. Occlusion training will help us providing unique beneficial training mode for promoting muscle hypertrophy. In control group players will perform general exercises session and in experimental sessions players will perform with occlusion training which is blood flow resistance training (BFR training shoulder, leg extension, bicep curls, kaatsu) 4 times a week for 4 weeks with 5 sets of 5 repetitions and then assessed pre-training and post-training values with assessment tools bench press, leg squat, leg power, maximum sprint time and pull-ups performed at 70% of 1-repetition maximum. This training will also improve and increase muscular strength in players.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Athletes with age group of 19-30 years of age.
* All players who had a minimum of two years of resistance training experience

Exclusion Criteria:

* Systemic issues with orthopedic issue, fractures, neuromuscular issue, cardiac issues.
* Players having history of prior surgery.

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
SQUATS | 4 weeks
  The squats test is a simple, yet effective way to monitor leg strength on a regular basis. To conduct this test a chair or box that makes the players knees bend at right angles when they are sitting. The players warm up for 10 minutes. Players stands in front of a chair, facing away from it, with their feet shoulder-width apart. The players squats down, lightly touching the chair with their backside before standing back up and repeats this sequence of movements until they are unable to continue.The assistant counts and records the number of completed squats.
BENCH PRESS | 4 WEEKS
  The objective of the bench press test is to evaluate an player's upper body strength. For bench press test for hockey players requirements are Barbell and weights, Weighing Scales and Bench. This test requires the athlete to complete as many bench presses as possible with no rest. The assistant weighs and records the athlete's weight. The players warm up for ten minutes .The assistant loads the barbell with a weight close to the players one repetition maximum load. The player conducts bench presses until they are unable to continue. The assistant acts as a spotter for the athlete and counts the number of successful bench presses. If the number of bench presses exceeds ten, then the athlete rests for ten minutes, the assistant increases the barbell weight, and the player repeats the test.
MAXIMUM TIME SPRINT | 4 WEEKS
  Sprints are used to primarily test an players acceleration. Max speed is directly linked to initial acceleration so testing sprint times at smaller initial intervals give a picture of whether training is improving acceleration and therefore max speed. This test involves a 40m sprint with 5m acceleration/deceleration spaces on either end of the test track. Timing lights are placed at 5m and 35m respectively. The players must complete 6 trials, with each trial beginning at 30-second intervals (0s, 30s, 60s, etc). Electronic timing gates are to be set up at the 0, 10, 30 and 40m marks Players start in a two-point standing stance, with the front foot in between the set of cones placed at the start line. 3 attempts are allowed. Players may remove themselves from testing once they feel they have given a maximal attempt. Data required: time for 10m, 30m, and 40m recorded to the nearest 0.01sec.
LEG POWER | 4 WEEKS
  The Power Index is a simple measure that is determined by calculating the square root of the athlete's body weight (in pounds) and multiplying it by the square root of their vertical jump (in inches). Drop Jump a test of leg strength and power which requires the athlete to drop off a box and immediately jump as high as they can. Standing Long (Broad) Jump Test: jump off two legs for maximal distance, a measure of leg power. The Vertical Jump Test can be performed to measure leg power.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No